CLINICAL TRIAL: NCT05628259
Title: The Effect of Tele-Nursing Based Motivational Interviewing on Diabetes Self-Efficacy, Diabetes Self-Management and Metabolic Control Parameters in Individuals With Type 2 Diabetes: Randomized Controlled Study
Brief Title: The Effect of Tele-Nursing Based Motivational Interviewing in Individuals With Type 2 Diabetes:RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Collaborators: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Principal Investigator, EDA KILINÇ İŞLEYEN, Assistant Profesor Dr., Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EKILINCISLEYEN
Record Dates: First submitted 2022-11-17; First posted 2022-11-28 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Type2 Diabetes; Self Efficacy; Self Management; Tele-nursing; Motivational Interview; LDL - Low Density Lipoprotein Receptor Disorder; High Density Lipoprotein Deficiency; Cholesterol; Lipidosis
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Hypoalphalipoproteinemias; Lipidoses

STUDY DESIGN:
Intervention Model Description: This study is a parallel group randomized controlled study.
Who Masked: Participant
Masking Description: Single blinding was provided that included inclusion criteria and agreement to participate in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A motivational interview (MI) program based on the telenursing approach was applied to the individuals in the experimental group. In this study, the MI procedure includes eight sessions in total, with four sessions of motivational interviews by phone in the first month of the intervention and four sessions of motivational interviews by phone in the next two months for each individual. Pre-tests were collected in the first month. Afterwards, MI intervention was applied for three months. This intervention was applied to the experimental group in addition to the routine care provided by the hospital. MI application took an average of 45-60 minutes via phone call.
  Interventions: Behavioral: Tele-Nursing based Motivational Interviewing
- Control Group (No Intervention): The control group received routine nursing care in the diabetes policlinic.

INTERVENTIONS:
Behavioral: Tele-Nursing based Motivational Interviewing — A motivational interview (MI) program based on the telenursing approach was applied to the individuals in the experimental group. In this study, the MI procedure includes eight sessions in total, with four sessions of motivational interviews by phone in the first month of the intervention and four sessions of motivational interviews by phone in the next two months for each individual. Pre-tests were collected in the first month. Afterwards, MI intervention was applied for three months. This intervention was applied to the experimental group in addition to the routine care provided by the hospital. MI application took an average of 45-60 minutes via phone call.
  Arms: Intervention Group

SUMMARY:
This study carried out to examine the effect of tele-nursing based motivational interviewing on diabetes self-efficacy, diabetes self-management and metabolic control parameters (Body mass index, waist circumference, HbA1c%,fasting blood glucose, LDL cholesterol, HDL cholesterol, total cholesterol, triglyceride) in individuals with type 2 diabetes.

DETAILED DESCRIPTION:
The first researcher of the article who applied Motivational Interviewing Techniques has a "Motivational Interviewing Techniques Training" certificate. A motivational interview (MI) program based on the telenursing approach was prepared by the researchers based on the literature for the individuals in the experimental group. In this study, the MI procedure includes eight sessions in total, with four sessions of motivational interviews by phone in the first month of the intervention and four sessions of motivational interviews by phone in the next two months for each individual. Pre-tests were collected in the first month. Afterwards, MI intervention was applied for three months. This intervention was applied to the experimental group in addition to the routine care provided by the hospital. MI application took an average of 45-60 minutes via phone call.

ELIGIBILITY:
Inclusion Criteria:

1) being over 18 years old, 2) receiving insulin or insulin + oral therapy, 3) diagnosis of type 2 diabetes at least one year ago, 4) having a BMI of 25 and above, 5) HbA1c value of 7 and above, 6) access to phone, 7) voluntarily agreeing to participate in the study.

Exclusion Criteria:

1) have a physical disability.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-10-02 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Efficacy Scale | Change from Baseline diabetes self-efficacy at 6 months
  The change in diabetes self efficacy of individuals with Type 2 diabetes at 3rd month and 6 rd month with the Diabetes Self-Efficacy Scale.
Diabetes Self-Management Scale | Change from Baseline diabetes self-management at 6 months
  This scale was used to measure the behavioral component of individuals in the IMB model. The validity and reliability study of the Turkish Diabetes Self-Management Perception Scale was conducted by Eroğlu and Sabuncu (2018). The scale consists of 16 items and 4 sub-dimensions and is a 4-point Likert type. Glucose Management sub-dimension: Items 4, 6, 10, 12 (items 4 and 12 are about drug use, items 1, 6 and 10 are about blood glucose monitoring). Diet Control sub-dimension: Items 2, 5, 9, 13. Physical Activity sub-dimension: Items 8, 11, 15. Use of Health Services sub-dimension: It consists of 3, 7, 14, and 16 items. The DMS scale consists of 16 items, 7 of which are straight and 9 of which are reversed. The scores of the items numbered "5, 7, 10, 11, 12, 13, 14, 15 and 16" in the scale are calculated by reversing them. Diabetes self-management increases as the score gets closer to 10.

SECONDARY OUTCOMES:
HbA1c% | Change from Baseline HbA1c% at 6 months
  Hemoglobin A1C
BMI | Change from Baseline Body Mass Index at 6 months
  Body Mass Index
FBG | Change from Baseline Fasting glucose at 6 months
  Fasting blood glucose
LDL | Change from Baseline LDL at 6 months
  Low-density lipoprotein
HDL | Change from Baseline HDL at 6 months
  High-density lipoprotein
waist circumference | Change from Baseline waist circumference at 6 months
  waist circumference
Total cholesterol | Change from Baseline total cholesterol at 6 months
  Total cholesterol
Triglyceride | Change from Baseline total triglyceride at 6 months
  triglyceride

CONTACTS AND LOCATIONS:
Overall Officials: Eda KILINÇ İŞLEYEN, PhD. RN., Study Chair — Uşak University
Locations (3):
- Turkey (Türkiye) (3):
  - Eda Kılınç İşleyen, Pamukkale, Denizli
  - İrem Nur ÖZDEMİR, Istanbul
  - Şengül AYDIN YOLDEMİR, Istanbul

REFERENCES:
- [Derived] Isleyen EK, Ozdemir IN, Yoldemir SA. The effect of tele-nursing based motivational interviewing on self-efficacy, self-management and metabolic control parameters in individuals with type 2 diabetes: randomized controlled study. Ir J Med Sci. 2025 Apr;194(2):563-573. doi: 10.1007/s11845-025-03916-5. Epub 2025 Feb 21. PMID 39982630